CLINICAL TRIAL: NCT01670461
Title: FAmily CEntered (FACE) Advance Care Planning for Teens With Cancer
Acronym: FACE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maureen Lyon (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor-Investigator, Maureen Lyon, Associate Research Professor in Pediatrics, Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PEP-10-171-01-PCSM
Record Dates: First submitted 2012-08-17; First posted 2012-08-22 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Cancer
Keywords: advance care planning, palliative care, pediatric
MeSH Terms: conditions — Neoplasms | interventions — Advance Care Planning; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FACE Advance Care Planning (Experimental): FACE intervention goal is to facilitate conversations about EOL care between adolescents and their legal guardians/surrogates to increase congruence in treatment preferences, to decrease decisional conflict, while supporting plans and actions, psychological adjustment and quality of life. Three 60 to 90-minute sessions in a dyadic format with a trained/certified interviewer. Session 1. The Lyon Family Centered Advance Care Planning Survey©. Session 2. Respecting Choices® Family-Centered Cancer Specific ACP Interview. Session 3. Completion of Five Wishes©.
  Interventions: Behavioral: FACE
- Standard of Care (SOC) Control (Other): Standard of Care Control: Advance Directive Information Booklet plus Advance Directive Checklist.
  Interventions: Behavioral: Standard of Care (SOC) Control

INTERVENTIONS:
Behavioral: FACE — FACE intervention goal is to facilitate conversations about EOL care between adolescents and their legal guardians/surrogates to increase congruence in treatment preferences, to decrease decisional conflict, while supporting plans and actions, psychological adjustment and quality of life. Three 60 to 90-minute sessions in a dyadic format with a trained/certified interviewer. Session 1. The Lyon Family Centered Advance Care Planning Survey©. Session 2. Respecting Choices® Family-Centered Cancer Specific ACP Interview. Session 3. Completion of Five Wishes©.
  Other Names: FAmily CEntered (FACE) Advance Care Planning
  Arms: FACE Advance Care Planning
Behavioral: Standard of Care (SOC) Control — Standard of Care (SOC) control will be provided with written information that encourages conversation the treatment team. At Children's National the following represent hospital policy: " … regarding advance directives … to honor each non-minor patient's wishes … to encourage and assist patients in determining and expressing their preferences regarding treatment decisions for use in the event they subsequently become unable to make such decisions." Upon admission if they do not have an advance directive, they should be given the "Advance Directive Information Booklet" and the Advance Directive Checklist. If they already have one, the patient is asked to provide a current copy, and it is placed in the medical record.
  Other Names: Standard of Care Control plus Information
  Arms: Standard of Care (SOC) Control

SUMMARY:
Advance Care Planning (ACP) prepares patients and their loved ones for future health care decisions, including end-of-life decisions. Yet, the needs of adolescent oncology patients for participation in ACP, despite its priority, is not well studied. Our goal is to test a model of ACP that anticipates these issues, fully empowers the family and adolescent, and keeps the key role of health care professionals central, building on our earlier work. We hypothesized FAmily CEntered (FACE) ACP, would: (1) increase congruence in treatment preferences between adolescents and surrogates; (2) decrease decisional conflict for adolescents; and (3) increase quality of communication compared with controls.

DETAILED DESCRIPTION:
Condition The purpose of the FACE intervention is to facilitate conversations about EOL care between adolescents and their legal guardians or surrogates in order to increase congruence in treatment preferences, to decrease decisional conflict, while supporting plans and actions, psychological adjustment and quality of life. This intervention will consist of three 60 to 90-minute sessions in a dyadic format with a trained/certified interviewer. Each session will be followed by a 15 minute assessment, using process measures to assess participants' ratings of the quality of the communication with the facilitator and satisfaction (negative and positive emotions in response to session) on a Likert scale. A research assistant, not the facilitator, will conduct the immediate post evaluation sessions. A Standard of Care comparison condition will also be assessed and measures administered at the same time intervals: at baseline, one week intervals for three weeks for process measures and Statement of Treatment Preferences, and at 3 month-post intervention follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥14.0 years and <21.0 years for adolescents at enrollment;
* Age ≥ 21.0 years for surrogates at enrollment;
* IQ > 70 or not known to be developmentally delayed;
* Depression score on Beck Depression Inventory, Second Edition (BDI-II) Total Score < 26;
* Primary language English

Exclusion Criteria:

* In foster care;
* Developmentally delayed;
* Suicidal or homicidal or psychotic at time of screening;
* Not understand or speak English; and
* Failure on mini mental status exam

Ages: 14 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Statement of Treatment Preferences | Week 3
  Statement of Treatment Preferences expresses values and goals related to future decision making regarding frequently occurring scenarios common to individuals dying of cancer). This instrument will be used to document specific treatment preferences of patients and the surrogate's understanding of what the patient would want. Patients and surrogates choose one of three options, "to continue all treatment and keep fighting," "to stop all treatment to prolong my life," and "don't know." It can also be used to monitor changes in patient's preferences over time. This tool has been used in adults and in adolescents in the FACE study conducted by the PI.

SECONDARY OUTCOMES:
Quality of Patient-Interviewer Communication | Week 2, 3 and 4
  Quality of Patient-Interviewer Communication is a questionnaire to be administered independently to patient and parent/surrogate following Sessions 1, 2 and 3, regardless of randomization. This tool will be used to evaluate the quality of communication that occurs between the patient/guardian/surrogate and the HCP/interviewer. This instrument consists of four items to determine the quality of patient-clinician communication. Items are rated on a 3-point scale with degree from "no" to "definitely yes," meaning that the higher scores indicate the higher satisfaction with the quality of communication. Good internal consistencies have been reported in patients with AIDS (Cronbach's α = .81.
Decisional Conflict Scale | Week 3
  Decisional Conflict Scale is used to measure the degree of uncertainty about the course of action to take. The DSC consists of three subscales on a five-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), e.g., "This decision was hard for me to make." The DSC demonstrated good test-retest item reliabilities (r≥.80).

OTHER OUTCOMES:
Beck Depression Inventory-II | Week 1 and Month 4 (plus or minus one month)
  Beck Depression Inventory-II (BDI-II)is a 21-item scale self-report measure to assess presence of symptoms of depression and severity of symptoms reported. This instrument has shown a high content, construct, and factorial validity and is appropriate for children and adolescents > 13 years of age. Reliability and validity are good.
Beck Anxiety Index (BAI). | Week 1 and Month 4 (plus or minus one month)
  Beck Anxiety Index (BAI). This is a 21-item measure assessing severity of subjective, somatic, and panic-related symptoms of anxiety. Participants rate the degree of discomfort experienced as a result of each symptom over the past week on a 4-point Likert scale (range 0-3). Items are summed with a maximum possible score of 63. Scores of 0 to 7 indicate minimal anxiety, 8-15 indicate mild anxiety, 16-25 indicated moderate anxiety, and >26 indicate severe anxiety. Test-retest reliability for this measure is acceptable (r = .75) as is internal consistency reliability (α = .92). The BAI has also demonstrated adequate content, concurrent, construct, discriminant, and factorial validity. This measure was validated to clinically assess severity of anxiety in individuals aged 17 to 80, however will be extended to the younger age range of this study to allow for consistency of data collected by a single measure of anxiety.
Five Wishes© | Week 4
  Five Wishes© (Towey, Aging with Dignity Component developed with support from The Robert Wood Johnson Foundation) is a legal document that facilitates having people express their treatment preferences if they were seriously ill or unable to communicate their wishes. The adolescent completed this along with their parent/proxy during the third experimental session. For adolescents under age 18, the Five Wishes© must be signed by their parent or legal guardian to be legally sufficient.
Threat Appraisal Scale (TAS). | Week 3
  Threat Appraisal Scale (TAS)is a questionnaire administered to the adolescent during baseline assessment only. This measure will retrospectively estimate the adolescent's threat appraisal of cancer when adolescent learned of cancer diagnosis. Test-retest reliability for this measure ranges from .68 in younger children to .93 in older children. TAS scores are found to demonstrate a high degree of agreement with children's open-ended descriptions of negative life events, indicating adequate convergent validity of this measure. Theoretically, threat appraisal is related to Lazarus' concept of primary appraisal, particularly to the way in which the event threatens the child's commitments, goals, or values. Higher threat appraisals should lead to negative arousal and coping and to increased psychological symptoms.
Spiritual Well Being Scale of the Functional Assessment of Chronic Illness Therapy - Version 4 (FACIT-Sp). | Week 1 and Month 4 (plus or minus one month)
  Spiritual Well Being Scale of the Functional Assessment of Chronic Illness Therapy - Version 4 (FACIT-Sp)is a questionnaire administered individually to both adolescent and guardian/surrogate. This measure will investigate spirituality as a protective process. This 23 item scale focuses primarily on the existential aspects of spirituality and faith. There are two subscales: meaning/peace and faith. The FACIT-SP has been used to study spirituality in teens with chronic illnesses.
The Pediatric Quality of Life Inventory™ 4.0 (PedQL™ 4.0) | Week 1 and Month 4 (plus or minus one month)
  The Pediatric Quality of Life Inventory™ 4.0 (PedQL™ 4.0). Adolescent and parent/surrogate will complete independently the age-appropriate self-report version and the parent proxy report version. This is a 23-item modular instrument designed to measure health-related quality of life (HRQOL) in children and adolescents. It measures four dimensions of functional quality of life (Core Scales: Physical, Emotional, Social, School) applicable to pediatric populations with acute and chronic health conditions. This measure was selected, because it has the strongest norms, validity, and reliability of the measures available.
Satisfaction Questionnaire | AWeek 2, 3 and 4
  The Satisfaction Questionnaire assesses negative and postive emotional reactions to participating in the study on the part of the adolescent and the surrogate decision-maker/family member. It was designed specifcally for this study based on community based participatory research.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen E Lyon, PhD, Principal Investigator — Children's Research Institute, Children's National Medical Center
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Lyon ME, Jacobs S, Briggs L, Cheng YI, Wang J. Family-centered advance care planning for teens with cancer. JAMA Pediatr. 2013 May;167(5):460-7. doi: 10.1001/jamapediatrics.2013.943. PMID 23479062
- [Result] Jacobs S, Perez J, Cheng YI, Sill A, Wang J, Lyon ME. Adolescent end of life preferences and congruence with their parents' preferences: results of a survey of adolescents with cancer. Pediatr Blood Cancer. 2015 Apr;62(4):710-4. doi: 10.1002/pbc.25358. Epub 2014 Dec 24. PMID 25545105
- [Result] Lyon ME, Jacobs S, Briggs L, Cheng YI, Wang J. A longitudinal, randomized, controlled trial of advance care planning for teens with cancer: anxiety, depression, quality of life, advance directives, spirituality. J Adolesc Health. 2014 Jun;54(6):710-7. doi: 10.1016/j.jadohealth.2013.10.206. Epub 2014 Jan 7. PMID 24411819
- [Result] Watson A, Weaver M, Jacobs S, Lyon ME. Interdisciplinary Communication: Documentation of Advance Care Planning and End-of-Life Care in Adolescents and Young Adults With Cancer. J Hosp Palliat Nurs. 2019 Jun;21(3):215-222. doi: 10.1097/NJH.0000000000000512. PMID 30829829